CLINICAL TRIAL: NCT01961856
Title: Platelet Reactivity After Ticagrelor Loading Dose Versus Clopidogrel Loading Dose and Reloading With Ticagrelor, in Patients With ST-elevation Myocardial Infarction (STEMI) Undergoing Primary Percutaneous Coronary Intervention (PCI).
Brief Title: Ticagrelor Loading Dose Versus Clopidogrel Loading and Reloading With Ticagrelor.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-17
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Platelet Reactivity
Keywords: platelet reactivity; ticagrelor loading dose; clopidogrel loading dose
MeSH Terms: interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Active Comparator): Ticagrelor 180mg loading dose
  Interventions: Drug: Ticagrelor
- Clopidogrel and Ticagrelor (Experimental): Clopidogrel 600mg loading dose followed by a Ticagrelor 180mg loading dose 2 hours later
  Interventions: Drug: Clopidogrel and Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel and Ticagrelor — Clopidogrel 600mg loading dose followed by Ticagrelor 180mg loading dose
  Arms: Clopidogrel and Ticagrelor
Drug: Ticagrelor — Ticagrelor 180mg loading dose
  Arms: Ticagrelor

SUMMARY:
In the PLATO substudy referring to patients presenting with an ST-elevation Myocardial Infarction(STEMI), out of the 4201 who received ticagrelor, 1326 had been pre-treated with a 600mg clopidogrel loading dose (LD) within 24 hours prior to randomization. It is a logical assumption, that patients who are being reloaded with ticagrelor will demonstrate reduced platelet reactivity (PR) at 24 hours, in comparison to those who were initially loaded with ticagrelor, due to the synergistic antiplatelet effect. Single loading with ticagrelor though, will possibly be accompanied by a smaller bleeding potency compared to reloading with ticagrelor. Therefore, we assume that single loading with ticagrelor is non-inferior to reloading with ticagrelor, in terms of platelet reactivity.

P2Y12 inhibitor naive patients with STEMI, they will be randomized immediately after coronary angiography (Hour 0) in receiving either Ticagrelor 180mg LD or Clopidogrel 600mg LD and 2 hours later reloading with Ticagrelor 180mg, after written informed consent. PR will be measured, using the VerifyNow assay at randomization (Hour 0) and at 2, 4, 6 and 24 hours post randomization. In addition, a 12-lead ECG will be performed before randomization, 90 and 180 minutes after the first balloon inflation, as well as on the exit day. Troponin I and CK-MB will be assessed at randomization and at hour 4, 12, 24, 48 and 72 after randomization.

Non inferiority of Ticagrelor LD versus Ticagrelor re-LD would be accepted if the upper bound of the 2-sided 95% CI around the estimated LS mean difference (Ticagrelor LD minus Ticagrelor re-LD) in the primary end point (PR at 24 hours) would lie bellow Δ=35 PRU. This non-inferiority margin (Δ) represents the upper bound of the LS mean difference in PR between Ticagrelor and Prasugrel arm at 24 hours after LD in a pharmacodynamic study of 55 STEMI patients.

Considering previous studies PR at 24 hours post randomization was estimated at 47±40 PRU and 41±35 PRU for Ticagrelor only LD and Ticagrelor re-LD group respectively. To obtain 85% statistical power with a 2-sided alpha=0.05, approximately 32 patients in each treatment group (64 in total) would be needed to establish the primary hypothesis using the abovementioned non-inferiority margin of 35 PRU. Anticipating a 5% dropout rate, enrollment was set to at least 68 patients. The primary endpoint, as well as PR at all the other time points of the study will be analyzed separately via a mixed effect model with treatment as fixed effect, patient as a random intercept and PR at baseline as a covariate. Least squares estimates of the mean difference will be presented, with 95% confidence intervals and a two-sided p-value for the treatment effect. P values for secondary endpoints will be reported for two-tailed tests of superiority.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Patients with STEMI (pain onset <12 hours) undergoing primary PCI
* P2Y12 inhibitor naive
* Written informed consent

Exclusion Criteria:

* Peri-procedural IΙb/IIIa inhibitor administration
* Cardiogenic shock/hemodynamic instability
* Pseudo-aneurism, retroperitoneal hematoma, major bleeding (need for transfusion or Hb decline≥5 gr/ dl)
* Need for anticoagulant treatment
* Current or future administration of other thienopyridines or ADP receptor inhibitors
* Known thrombocytopenia (<100.000 / μL) at randomization
* Hct <30% or Hct > 52% during randomization
* Known allergy to clopidogrel or ticagrelor
* Recent (< 6 weeks) major operation, including CABG
* History of bleeding disorders
* Known intracranial mass, arteriovenous shunt or aneurism
* Previous intracranial bleeding
* INR>1,5
* Other clinical conditions associated with increased bleeding risk, according to the investigators' judgment
* Known creatinine Clearance <30ml/h at randomization or hemodialysis
* Severe/moderate liver failure
* Pregnancy/ breastfeeding
* Increased risk for bradyarrhythmias, according to the investigator's judgment
* Administration of potent CYP3A inhibitor (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, grapefruit juice N1 L/d), substrates of CYP3A with narrow therapeutic range (cyclosporine, quinidine), or potent CYP3A inducers (rifampin /rifampicin, phenytoin, carbamazepine)
* Severe uncontrolled chronic obstructive pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Platelet Reactivity between the two groups at 24 hours | 24 hours

SECONDARY OUTCOMES:
Platelet reactivity between the two groups at 4 hours | 4 hours

OTHER OUTCOMES:
Platelet reactivity between the two groups at hour 2 | 2 hours
Percentage of patients presenting high platelet reactivity (HPR) (≥208 PRU) between the two groups at hour 2 | 2 hours
Percentage of patients presenting high platelet reactivity (HPR) (≥208 PRU) between the two groups at hour 4 | 4 hours
Percentage of patients presenting high platelet reactivity (HPR) (≥208 PRU) between the two groups at hour 6 | 6 hours
Percentage of patients presenting high platelet reactivity (HPR) (≥208 PRU) between the two groups at hour 24 | 24 hours
Overall ST segment deviation in all electrocardiogram leads except aVR between groups at 90 min after first balloon inflation | 90 min
Overall ST segment deviation in all electrocardiogram leads except aVR between groups at 180 minutes after the first balloon inflation | 180 minutes
Overall ST segment deviation in all electrocardiogram leads except aVR between groups at discharge | 5 days
Percentage of patients with ≥50% resolution of ST deviation in all leads except aVR (in comparison to hour 0) at 90 minutes after the first balloon inflation, between the two groups. | 90 minutes
Percentage of patients with ≥50% resolution of ST deviation in all leads except aVR (in comparison to hour 0) at 180 minutes after the first balloon inflation, between the two groups. | 180 minutes
Percentage of patients with ≥50% resolution of ST deviation in all leads except aVR (in comparison to hour 0)at discharge, between the two groups. | 5 days
Percentage of patients with ≥50% resolution of ST elevation in all leads except aVR (in comparison to hour 0) at 90 minutes after the first balloon inflation, between the two groups. | 90 minutes
Percentage of patients with ≥50% resolution of ST elevation in all leads except aVR (in comparison to hour 0) at 180 minutes after the first balloon inflation, between the two groups. | 180 minutes
Percentage of patients with ≥50% resolution of ST elevation in all leads except aVR (in comparison to hour 0) at discharge between the two groups. | 5 days
Overall ST segment elevation in all electrocardiogram leads except aVR between groups at 90 min after first balloon inflation | 90 minutes
Overall ST segment elevation in all electrocardiogram leads except aVR between groups at 180 min after first balloon inflation | 180 min
Overall ST segment elevation in all electrocardiogram leads except aVR between groups at discharge | 5 days
Area under the curve (AUC) defined by Troponin I values assessed at 0 hour, 4, 12, 24, 48 and 72 hours between the two groups. | 72 hours
Area under the curve (AUC) defined by CK-MB values assessed at 0 hour, 4, 12, 24, 48 and 72 hours between the two groups. | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Patras University Hospital, Pátrai, Achaia, Greece